CLINICAL TRIAL: NCT04139538
Title: Changes of Oral Microbiome and Immunogenity of Saliva During Orthodontic Therapy With Aligners and Multibracket Therapy - a Pilot Study
Brief Title: Microbiome and Immunogenity of Saliva During Orthodontic Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Michael Nemec, Staff member, dentist, Medical University of Vienna
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: 1288/2019
Record Dates: First submitted 2019-09-22; First posted 2019-10-25 (Actual); Last update posted 2023-03-23 (Actual); Status verified 2023-03

CONDITIONS: Orthodontic Appliances, Removable; Orthodontic Appliances, Fixed; Oral Microbiome; Cell Culture; Periodontal Index
MeSH Terms: interventions — Orthodontics

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Invisalign treatment (Experimental): Aligner patients will be treated with Invisalign® aligners to correct malocclusion
  Interventions: Procedure: orthodontic treatment
- selfligating bracket treatment (Active Comparator): Multibracket patients will be treated with self ligating orthodontic brackets
  Interventions: Procedure: orthodontic treatment

INTERVENTIONS:
Procedure: orthodontic treatment — Malocclusion will be treated with orthodontic appliances (fixed or removable)

SUMMARY:
There are two essential ways of treatment in the field of orthodontics. The fixed appliance treatment with self-ligating or conventional brackets and treatment with aligners. Fixed orthodontic treatment has been the optional therapy for decades. Due to an increasing demand of patients for a more aesthetic treatment, the number of aligner treatments multiplied over the last years. Within the last years, a crucial role of oral microbiome in the maintenance of oral health was largely appreciated. However, to date there is no data on the effect of different orthodontic treatments on the oral microbiome. The aim of the research project is the prospective comparison of the oral microbiome in saliva of adult patients treated with Invisalign® aligners or metal brackets. We plan to include a sample of twenty healthy individuals. Half of the participants will receive aligner treatment with Invisalign® and half metal brackets. Saliva will be collected before, 3 and 6 months after the beginning of the orthodontic therapy via a stimulated a saliva collection. The 16S rDNA genes will be amplified and sequenced with Illumina MiSeq® System. Probing depth, bleeding on probing and Plaque Index will be evaluated over time and correlated with changes of the oral microbiome.

DETAILED DESCRIPTION:
Adult patients (18 years and older) from the Clinical Division of Orthodontics at the University Clinic of Dentistry Vienna will be invited to participate in this pilot microbiologic study according to defined inclusion/exclusion criteria after giving their consent. This study is a pilot project and therefore no sample size calculation will be made. Twenty patients will be treated with Invisalign® aligners and twenty patients will receive multibracket therapy. A previous microbiological study showed that lingual orthodontic therapy has a short-term effect on oral microflora. Another microbial study on colonization on dental implants also reported bacterial shift upon implant therapy.

All patients will get instructions in oral hygiene on the day when clinical records are gathered. On the day when the treatment plan will be presented to the patient, the Plaque Index will be evaluated by a trained orthodontist. For the start of the treatment a Plaque Index of < 20% is required. On the day before the orthodontic treatment is started, T0 sample collection will be conducted and periodontal indices will be assessed. A clinical examination including periodontal probing depth, bleeding on probing, and Plaque Index (PI) will be performed before (T0), after 3 months (T1) and after 6 months of the beginning of either aligner or bracket therapy. Microbiological sampling will be performed by stimulated saliva collection according to our protocol. Saliva samples will be divided in aliquots in stored in cryo-tubes at -80°C. Molecular detection of microorganisms by sequencing of 16S rDNA genes, sequencing analysis and taxonomic assignment will be performed at the Department of Laboratory Medicine at the Medical University of Vienna.

By sequencing of 16s rDNA genes with sequencing analysis and taxonomic assignment of bacteria in saliva we expect to reveal possible shifts in microbial phyla/genera between various time points. Metagenomic studies are commonly performed by analysing the prokaryotic 16S ribosomal RNA gene (16S rRNA), which is approximately 1,500 base pairs long and contains nine variable regions interspersed between conserved regions. Variable regions of 16S rRNA are frequently used in phylogenetic classifications such as genus or species in diverse microbial populations.

DNA Extraction:

Due to better quantitative and qualitative results in comparison to commercial DNA extraction kits, DNA will be isolated with a modified CTAB SDS chloroform-based method. Mechanical analysis will be carried out using 1mm silica spheres under addition of proteinase K (Qiagen, Venlo, Netherlands) as well as the detergents SDS (sodium dodecyl sulfate) and CTAB (cetyltrimethylammonium bromide). After extraction, the DNA quantity will be determined with Qubit® 2.0 via the dsDNA HS kit (Life Technologies, Carlsbad, California) and NanoDrop 2000c spectrophotometer (Thermo Scientific, Waltham, Massachusetts). Additionally, the absorption ratios A260/280 and A260/230 will be used to estimate the purity of the DNA.

Metagenome Analysis:

The overall composition of the bacterial organisms in the samples will be evaluated by analysing microbiome. Therefore, we will use high throughput sequencing with the MiSeq® platform (Illumina, San Diego, California). We will analyse the variable V3 and V4 regions of the 16S rRNA gene. For the phylogenetic classification, the bacterial 16S rRNA will be amplified using primers 27F (5'-CCT ACG GGN GGC WGC AG-3') and 1391R (5'-GACTACHVGGGTATCTAATCC-3').

Bioinformatic analysis:

The quality of the Next Generation Sequencing run will be assessed using the software FASTQC 0.11.4. The removal of low-quality bases will be carried out with the Trimmomatic-0.35 software . For sequence analysis and clustering similar sequences into clusters (OTUs) the UPARSE pipeline will be utilized. For comparison and statistical analysis of the microbiome data we will use RStudio (Team 2016) as platform with R as language (R Development Core Team 2010) and different R-packages.

ELIGIBILITY:
Inclusion Criteria:

* Class I skeletal relationship
* Normo-divergent Frankfort Mandibular-Plane Angle
* Minimal mandibular crowding in range from 1 to 3 according to Little's Index (Little 1975)

Exclusion Criteria:

* Smoking habit
* Presence of extensive dental restorations in proximity to the gingival margin
* Presence of fixed bridges/crowns or partial dentures
* Previous periodontal nonsurgical treatment (such as full mouth disinfection, quadrant-by-quadrant therapy, full mouth debridement) within the past year
* Medications such as antibiotics, steroids, or nonsteroidal anti-inflammatory drugs within the past 6 months.
* Plaque Index > 20% before start of treatment Diabetes Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2022-09-01 (Actual); Study Completion 2024-10-01 (Estimated)

PRIMARY OUTCOMES:
changes of oral microbiome | up to 6 months
  bacteria of the oral microbiome including cariogenic bacteria via dna sequencing
changes of periodontal parameters | up to 6 months
  plaque index
changes of periodontal parameters | up to 6 months
  probing depth
changes of periodontal parameters | up to 6 months
  bleeding on probing

SECONDARY OUTCOMES:
immunogenity of saliva on oral cells in vitro | up to 2 weeks
  changes in viability
immunogenity of saliva on oral cells in vitro | up to 2 weeks
  gene expression changes via PCR

CONTACTS AND LOCATIONS:
Locations (1):
- Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Klindworth A, Pruesse E, Schweer T, Peplies J, Quast C, Horn M, Glockner FO. Evaluation of general 16S ribosomal RNA gene PCR primers for classical and next-generation sequencing-based diversity studies. Nucleic Acids Res. 2013 Jan 7;41(1):e1. doi: 10.1093/nar/gks808. Epub 2012 Aug 28. PMID 22933715
- [Background] Edgar RC. UPARSE: highly accurate OTU sequences from microbial amplicon reads. Nat Methods. 2013 Oct;10(10):996-8. doi: 10.1038/nmeth.2604. Epub 2013 Aug 18. PMID 23955772
- [Background] Levrini L, Mangano A, Montanari P, Margherini S, Caprioglio A, Abbate GM. Periodontal health status in patients treated with the Invisalign((R)) system and fixed orthodontic appliances: A 3 months clinical and microbiological evaluation. Eur J Dent. 2015 Jul-Sep;9(3):404-410. doi: 10.4103/1305-7456.163218. PMID 26430371
- [Background] Demling A, Demling C, Schwestka-Polly R, Stiesch M, Heuer W. Short-term influence of lingual orthodontic therapy on microbial parameters and periodontal status. A preliminary study. Angle Orthod. 2010 May;80(3):480-4. doi: 10.2319/061109-330.1. PMID 20050740
- [Background] de Freitas AR, Silva TSO, Ribeiro RF, de Albuquerque Junior RF, Pedrazzi V, do Nascimento C. Oral bacterial colonization on dental implants restored with titanium or zirconia abutments: 6-month follow-up. Clin Oral Investig. 2018 Jul;22(6):2335-2343. doi: 10.1007/s00784-018-2334-0. Epub 2018 Jan 18. PMID 29349504
- [Background] Haririan H, Andrukhov O, Bertl K, Lettner S, Kierstein S, Moritz A, Rausch-Fan X. Microbial analysis of subgingival plaque samples compared to that of whole saliva in patients with periodontitis. J Periodontol. 2014 Jun;85(6):819-28. doi: 10.1902/jop.2013.130306. Epub 2013 Oct 21. PMID 24144271
- [Background] Ren Y, Vissink A. Cytokines in crevicular fluid and orthodontic tooth movement. Eur J Oral Sci. 2008 Apr;116(2):89-97. doi: 10.1111/j.1600-0722.2007.00511.x. PMID 18353001